CLINICAL TRIAL: NCT04412265
Title: Relationship Between Frailty and Clinical Outcomes in Elderly Patients With COVID-19
Brief Title: Frailty in Elderly Patients With COVID-19
Acronym: FRA-COVID
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: FRA-COVID
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: Coronavirus; sars-covid-2; coronavirus infection; geriatrics
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid 19 patients: The study will be conducted on all patients hospitalized affected by pneumonia COVID related.
  Interventions: Other: Relation between frailty and clinical outcomes in elderly patients with COVID-19.

INTERVENTIONS:
Other: Relation between frailty and clinical outcomes in elderly patients with COVID-19. — To evaluate whether a tool built to measure frailty in elderly patients hospitalized in COVID + hospital departments are more accurate in predicting clinical outcomes compared to a clinical evaluation based on age and comorbidity. If the assessment of fragility were actually more accurate, the tool developed could be implemented in hospitals to support the clinician 's choices regarding the "roof of care" and actions to be taken undertake to prevent deterioration.

SUMMARY:
This is a multicentric retro-prospective observational study that wants to evaluate the relation between frailty and clinical outcomes in elderly patients with COVID-19.

DETAILED DESCRIPTION:
BACKGROUND:

Assessment of frailty is today the best way to evaluate the biological age of the elderly person. Fragility can be defined as a syndrome selected by the reduction of organized reserves and by the decreased resistance to "stressors", resulting from the cumulative decline of multiple physiological systems that cause vulnerabilities and adverse consequences.

The impact of fragility on clinical outcomes has been investigated in numerous studies conducted on elderly patients in various care setting, proving in all of them a significant and more reliable predictor of variables such as age, comorbidity and individual pathologies, short and long-term mortality, length of stay and the onset of complications.

Previous studies have already shown that frail older adults have a greater susceptibility to viral infections (including non-COVID-19 coronavirus) due to a malfunction of their immune system.

The identification of fragility could therefore be particularly useful for identifying subjects at risk of negative outcomes (worsening of respiratory parameters, need for intubation, mortality) even in a ward with COVID + patients. In other words, the imperceptible clinical heterogeneity behind the age parameter could be better represented by a multidimensional parameter capable of measuring the accumulation of age-related deficits.

SAMPLE SIZE (n. patients):

The study plans to recruit 30 subjects per week on average; for an expected total of about 300 subjects for each participating site.

STUDY DESIGN:

The patient will be enrolled in the study when obtaining consent. In this phase the following data will be collected:

* date of birth
* gender
* demographic data
* comorbidity
* Brescia_COVID respiratory scale
* modified Early Warning Score
* delirium
* data relating to functional autonomy
* blood chemistry data at the entrance.

Using the variables that are part of the Comprehensive Geriatric Assessment, it will be possible to calculate the Frailty Index (FI), according to the Rockwood deficit accumulation model. A series of variables will then be collected relating to treatment procedures, therapies, the team's choice to maximize the care ceiling for the individual patient and the patient's clinical outcome.

Patients will be treated as per Normal Clinical Practice; no blood chemistry tests will be required in addition to the panel of tests provided by the hospital's health management for all patients with COVID-19.

Given the difficulty in systematically obtaining written informed consent and given the great public interest of the project, the research will be conducted in the context of the authorizations guaranteed by Article 89 of the GDPR EU Regulation 2016/679, which guarantees the treatment for purposes of public interest, scientific or historical research or statistical purposes of health data.

STATISTICAL ANALYSIS:

The FI will be built according to the Rockwood deficit accumulation model, taking into account a minimum number of variables that are part of the Comprehensive Geriatric Assessment. The FI will be obtained from the ratio between the number of pathological conditions present and the total number of indicators evaluated. Data from patients older than 60 years of age will be compared.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of COVID related pneumonia
* Informed consent freely granted

Exclusion criteria

- Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on all patients hospitalized in COVID+ departments of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 1344 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Development of a tool to measure frailty | Until patient discharge from the hospital (approximately 1 year).
  The aim of the project is to evaluate whether a tool built to measure frailty in elderly patients admitted to the COVID + hospital wards is more accurate in predicting clinical states than a clinical evaluation developed on age and comorbidity.

SECONDARY OUTCOMES:
A "proxy" variable of the fragility index can be built on the basis of regional administrative databases only. | Until patient discharge from the hospital (approximately 1 year).
  Assess whether a "proxy" variable of the fragility index can be built on the basis of regional administrative databases only, which is able to predict the clinical outcomes of COVID + patients better than age and comorbidities alone.
Give elements to focus the screening policies for COVID19. | Until patient discharge from the hospital (approximately 1 year).
  Relate different levels of chronicity with the susceptibility of the elderly subject to infection to give elements to focus the screening policies for COVID19.
Give the prevention of contagion at the elderly population level. | Until patient discharge from the hospital (approximately 1 year).
  Relate different levels of chronicity with the susceptibility of the elderly subject to infection to prevent the contagion at the elderly population level.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Dipartimento di Geriatria, Fondazione Poliambulanza, Brescia
  - Dipartimento di Medicina e Riabilitazione, Istituto Clinico Ospedale S. Anna, Brescia
  - UO Malattie Infettive, Spedali Civili, Brescia
  - UOC Medicina I a indirizzo Geriatrico, Spedali Civili, Montichiari
  - ASST Monza-Ospedale San Gerardo, Monza
  - SCDU Geriatria, AOU Città della Salute e della Scienza - Presidio Molinette, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Johnstone J, Parsons R, Botelho F, Millar J, McNeil S, Fulop T, McElhaney J, Andrew MK, Walter SD, Devereaux PJ, Malekesmaeili M, Brinkman RR, Mahony J, Bramson J, Loeb M. Immune biomarkers predictive of respiratory viral infection in elderly nursing home residents. PLoS One. 2014 Oct 2;9(9):e108481. doi: 10.1371/journal.pone.0108481. eCollection 2014. PMID 25275464
- [Background] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Derived] Trevisan C, Grande G, Rebora P, Zucchelli A, Valsecchi MG, Foca E, Ecarnot F, Marengoni A, Bellelli G. Early Onset Delirium During Hospitalization Increases In-Hospital and Postdischarge Mortality in COVID-19 Patients: A Multicenter Prospective Study. J Clin Psychiatry. 2023 Aug 21;84(5):22m14565. doi: 10.4088/JCP.22m14565. PMID 37616485